CLINICAL TRIAL: NCT05214365
Title: Physiological Pacing vs.Conventional Pacing in the Prevention of Pacemaker-induced Cardiomyopathy: A Randomized Study
Brief Title: Physiological Pacing for AV Block to Prevent Pacemaker-induced Cardiomyopathy
Acronym: PHYSPAVB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Centro de Investigación Biomédica en Red Enfermedades Cardiovasculares (CIBERCV) (Unknown)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Head of Arrhythmia Section. Professor of Cardiology, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHYSPAVB
Record Dates: First submitted 2022-01-17; First posted 2022-01-28 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Conduction System Pacing; Conventional Ventricular Pacing
Keywords: Pacemaker-induced cardiomyopathy

STUDY DESIGN:
Intervention Model Description: Randomized, unicentric, simple blind.
Who Masked: Participant
Masking Description: The patient will be explained to be randomized to either one of the two branches. The type of therapy applied will not be communicated to the patient. The follow-up will be the same in the two branches. During the visits it will not be said which therapy has been applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional stimulation (Active Comparator): An electrode (in the apical or septal portion) will be implanted at the discretion of the implanter physician. Parameters of (sensing, impedance and threshold) will be measured as is usually done in our center.
  Interventions: Device: Pacemaker implantation and conventional cardiac pacing
- Physiological stimulation (Active Comparator): Pacing the his-purkinje system.
  Interventions: Device: Conduction system pacing implant

INTERVENTIONS:
Device: Pacemaker implantation and conventional cardiac pacing — Patients will have the pacemaker implanted in the electrophysiology laboratory. Electrode will be implanted (in the apical or septal portion) according to the criteria of the implanting physician.
  Arms: Conventional stimulation
Device: Conduction system pacing implant — Right ventricular lead was placed to get his bundle or left bundle branch.
  Arms: Physiological stimulation

SUMMARY:
The implantation of a pacemaker and conventional cardiac pacing from the right ventricle (apex or septum) is an effective and safe therapy for the treatment of patients with atrioventricular block and bradycardia.

DETAILED DESCRIPTION:
Pacemaker implantation and conventional cardiac stimulation from the right ventricle is an effective and safe therapy for the treatment of patients with atrioventricular block and bradycardia. But it can cause worsening of heart function, with a significant drop in LV ejection fraction, known as pacemaker-induced cardiomyopathy (PICM).

Conduction system pacing (either by his or left bundle branch pacing) causes a physiological left ventricular activation through the normal conduction system thus correcting the electrical and mechanical asynchrony caused by conventional pacing. Conduction system pacing may prevent the appareance of PICM.

Clinical, electrocardiographic, echocardiographic follow-up will be performed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥ 18 years of age.
* The patient must indicate their acceptance to participate in the study by signing an informed consent document.
* Patients with EF> 50% and indication for pacemaker implantation due to atrial-ventricular block according to current clinical guidelines.

Exclusion Criteria:

* Inability to understand and sign the informed consent.
* Patients with severe comorbidities and life expectancy <1 year.
* Patients with severe cognitive impairment or other comorbidities resulting in dependence for basic activities of daily life.
* Patients who cannot come to our center to carry out the follow-up of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Compare the incidence of pacemaker-induced heart disease | 12 months
  Pacemaker induced cardiomyopathy defined as appearance of ventricular dysfunction LVEF <45% or admission due to heart failure.

SECONDARY OUTCOMES:
Change in end-systolic volume. | 12 Months
  VTSVI
Correction of septal flash. | 12 Months
  Correction of septal flash determined with echocardiography (M mode)
Incidence of new onset of atrial fibrillation. | 12 Months
Hospitalization due to heart failure. | 12 Months
  Hospitalization: patient hospitalization (yes/no)
New York Heart Association functional classification. | 12 Months
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Pacing thresholds. | 12 Months
  Pacing thresholds.
Total implantation and electrode implantation times. | 12 Months
  Total implantation and electrode implantation times.
Adverse events. | 12 Months
  Resulted in reintervention or the termination of significant device function
Six minute walking test. | 12 Months
  Six minute walking test.
The Quality of Life Scale. | 12 Months
  The Minnesota living with heart failure questionnaire. The most widely used health-related quality of life questionnaires for patients with heart failure. Values from 0 to 105 (more is worse).
NT-proBNP. | 12 Months
  NT-proBNP measure

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Tolosana, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; Lluís Mont, MD, PhD, Study Director — Hospital Clinic of Barcelona; Margarida Pujol Lopez, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No